CLINICAL TRIAL: NCT02795455
Title: Reward Systems and Food Avoidance in Adolescents With Low Weight Eating Disorders
Brief Title: Reward Systems and Food Avoidance in Eating Disorders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Tom Hildebrandt, Associate Professor - Psychiatry, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GCO 15-0939; 1R01MH109639-01A1 (NIH)
Record Dates: First submitted 2016-05-19; First posted 2016-06-10 (Estimated); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Low Weight Eating Disorders; Anorexia Nervosa
Keywords: Eating Disorders; Food Avoidance; Reward Learning; Reward System; Family-based treatment; interoceptive exposure; insula-amygdala-ventral striatum subcircuits
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Interoceptive Exposure (IE) (Experimental): IE is an exposure-based intervention that involves consuming a food in session and tolerating uncomfortable feelings around eating.
  Interventions: Behavioral: Interoceptive Exposure (IE); Dietary Supplement: meal replacement shake
- Family Based Therapy-Weight Gain Control (FBT-WG) (Active Comparator): Family-based therapy uses parent(s) to help modify disordered eating and develop contingencies to motivate eating.
  Interventions: Behavioral: Family Based Therapy-Weight Gain Control (FBT-WG)
- Healthy Controls (HC) (No Intervention): HC participants will only participate in the pre and post-intervention visits and not in the intervention sessions.

INTERVENTIONS:
Behavioral: Interoceptive Exposure (IE) — Participants are provided with a meal replacement shake of 'unknown' Kcal or macronutrient content and are asked to mindfully observe the sensations (aversive taste, texture, bloating, icky feeling, etc.) and associated emotional states (i.e., disgust) with the empathetic support of parents/therapist in session, without expectation of habituation. Sessions occur on a weekly basis with session one lasting 2 hrs. The remaining 5 sessions last one hour, and participants eat a meal replacement shake over 30-minutes, identical to the first session. All sessions include debriefing and development of IE homework that includes daily practice of IE.
  Arms: Interoceptive Exposure (IE)
Behavioral: Family Based Therapy-Weight Gain Control (FBT-WG) — Participants and families randomized to FBT-WG will receive 6-weeks of FBT treatment for AN. Sessions occur weekly, with the first session lasting two hours and the remaining 5 sessions one hour. FBT is atheoretical in terms of the etiology, but uses parent-enforced contingencies to increase value of eating and decrease the value of food avoidance.
  Arms: Family Based Therapy-Weight Gain Control (FBT-WG)
Dietary Supplement: meal replacement shake
  Arms: Interoceptive Exposure (IE)

SUMMARY:
The researchers plan to explore brain networks involved in emotion processing and learning using a brain scan and test meals. One core feature of Anorexia Nervosa (AN) is eating a small number of high-calorie or high-fat foods. By studying why individuals with AN are disgusted by food or other eating situations, the researchers will be able to understand more about the neurobiological pathways that lead to restricting food intake and food avoidance. This study also aims to find whether one of two short-term interventions (Interoceptive Exposure (IE); Family-Based Therapy (FBT)) affects connections in the brain and if the treatments affect food avoidance. IE is an intervention that helps reduce anxiety about eating. FBT is an intervention that motivates patients to eat through working with family to increase the value of eating and decrease the value of avoiding foods.

DETAILED DESCRIPTION:
Anorexia nervosa (AN), a characteristically relentless pursuit of thinness with an intense fear of weight gain despite significantly low body weight, is a serious psychiatric disorder with high rates of morbidity and mortality. Low weight eating disorders (LW-ED), the broader category of eating pathology that includes AN and similar variants, are characterized by a chronic course, poor response to treatment, and food avoidance. Emerging neuroimaging evidence suggests that deficits in insula-amygdala-ventral striatum (IAVS) neurocircuitry contribute to individual variability in aversive and reward learning, and that these brain regions demonstrate abnormal responses to food/eating stimuli. The researchers' pilot data suggest that patients with LW-ED experience difficulty extinguishing food-cue associations in a reversal learning paradigm compared to healthy controls, a difficulty that is related to psychophysiological measures of aversive disgust (not fear). The researchers have also successfully piloted an interoceptive exposure intervention for this population that targets visceral sensitivity and seeks to increase 'top-down' regulation of the IAVS neurocircuit. The proposed project will (a) use novel fMRI-EMG to test the relationship between effective connectivity within amygdala-insula-ventral striatum network and its relationship to psychophysiological and behavioral measures of acute threat and reward learning in 60 adolescents with LWEDs and 30 healthy controls, (b) test the sensitivity of this network to an experimental interoceptive exposure paradigm relative to patients receiving family based therapy for weight restoration using dynamic causal modeling of fMRI-EMG data pre-post experimental conditions, (c) validate this model against objective measures of laboratory and real world eating behavior. The results of this study will help better understand the core neurocircuitry that underlies both threat processing and reward/aversive learning and how this circuit relates to objective behavior. Further, the researchers will determine the modifiability of this neurocircuitry via two distinct behavioral interventions chosen to target different aspects of affective processing and reward learning. These data will be used to inform future clinical interventions targeting aversive/reward learning within this population and dysregulation in insula-amygdala-ventral striatum subcircuits.

ELIGIBILITY:
Low Weight ED Patients

Inclusion criteria:

* Females,
* Adolescents ages 12-18,
* Speak English,
* Seeking treatment
* Refusal to maintain greater than minimally low body weight based on BMI for age percentiles and growth trajectories,
* Clinically significant restriction of food intake on the dietary restraint subscale of the EDE or evidence of persistent food avoidance as reported by patient or guardians.
* Given medical clearance from pediatrician or equivalent.

Exclusion criteria:

* Current psychotropic medication that would have an effect on performance on behavioral tasks (i.e., anti-anxiety medication),
* Comorbid psychotic or bipolar disorder,
* Active suicidal ideation,
* Major medical illness known to influence eating or weight,
* Current substance dependence,
* Previous exposure therapy for LW-ED.
* Physical limitation that would prevent participation (e.g., allergic to chocolate),
* For patients with current or a history of sexual or physical abuse by parents, siblings, or guardians, perpetrators of the abuse will be excluded from treatment; if physical or sexual abuse by a family member occurs during the course of treatment, perpetrators will be excluded from ongoing treatment

Healthy Comparison Adolescents

Inclusion criteria:

* Females,
* Adolescents ages 12-18,
* Speak English.

Exclusion criteria:

* Current psychotropic medication that would have an effect on performance on behavioral tasks (i.e., stimulant medication),
* Current or lifetime history of any psychiatric disorder, including eating disorders by K-SADS,
* Current or lifetime history of learning disorder or developmental disability
* Active suicidal ideation,
* Major medical illness,
* Other physical limitation that would prevent participation (e.g., allergic to chocolate).

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 90 (Actual)
Dates: Start 2016-11; Primary Completion 2021-07-29 (Actual); Study Completion 2021-07-29 (Actual)

PRIMARY OUTCOMES:
fMRI-EMG | Baseline and 6 weeks
  Change in the emotional responses from facial muscle movements to food pictures and non-food pictures as measured with the fMRI-EMG.

SECONDARY OUTCOMES:
KCal Intake | Baseline and 6 weeks
  Change in KCal Intake at 6 weeks as compared to baseline. Consumption of a standardized strawberry yogurt shake test meal will be measured in kcal. Participants will be presented with an 83 fluid ounce (2454.60-mL) covered opaque container containing approximately 1500 grams (1.04 kcal per gram, or approximately 1560 kcal) of strawberry yogurt shake. Patients will be informed that the meal consists of a strawberry yogurt shake, but will not be told the amount provided in the container. The instructions will direct participants to consume as much of the shake as they would like and that the meal will serve as their lunch (or dinner) for the day and to avoid touching or manipulating the container in any way.
Eating Disorder Examination (EDE) | Baseline and 6 weeks
  Change in EDE at 6 weeks as compared to baseline. Clinical interview to assess for eating disorder symptomology.
Clinical Impairment Assessment | Baseline and 6 weeks
  Change in assessment at 6 weeks as compared to baseline. The Clinical Impairment Assessment (CIA) is a 16-item self-report measure of the severity of psychosocial impairment due to eating disorder features on the past 28 days. Each item are scored 0, 1, 2, 3 with a higher rating indicating a higher level of impairment, with total score ranging from 0 to 48 with a higher score being indicative of a higher level of psychosocial impairment secondary to eating disorder features.
Anxiety Sensitivity Index-III | Baseline and 6 weeks
  Change in index at 6 weeks as compared to baseline. Self-reported anxiety symptomology

CONTACTS AND LOCATIONS:
Overall Officials: Tom Hildebrandt, PsyD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schulz KP, Sysko R, Fan J, Hildebrandt TB. Interoceptive Exposure Impacts Food-Cue Extinction in Adolescents With Low-Weight Eating Disorders: A Functional Magnetic Resonance Imaging Study. J Am Acad Child Adolesc Psychiatry. 2026 Jan;65(1):66-75. doi: 10.1016/j.jaac.2024.12.013. Epub 2025 Feb 25. PMID 40015474
- [Derived] Hildebrandt T, Schulz K, Fleysher L, Griffen T, Heywood A, Sysko R. Development of a methodology to combine fMRI and EMG to measure emotional responses in patients with anorexia nervosa. Int J Eat Disord. 2018 Jul;51(7):722-729. doi: 10.1002/eat.22893. Epub 2018 Aug 18. PMID 30120839

DOCUMENTS (2):
  • Study Protocol (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT02795455/Prot_000.pdf
  • Statistical Analysis Plan (2022-04-12): https://cdn.clinicaltrials.gov/large-docs/55/NCT02795455/SAP_001.pdf